CLINICAL TRIAL: NCT01861119
Title: Silicone Gel Versus Onion Extract Gel as Prevention for Postsurgical Scars: a Randomized Controlled Trial
Brief Title: Silicone Gel Versus Onion Extract Gel as Prevention for Postsurgical Scars
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CHA University (Other)
Responsible Party: Principal Investigator, Taejong Song, Professor, CHA University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: KNC13-020
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Hypertrophic or Keloid Scars
MeSH Terms: conditions — Hypertrophy; Keloid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Silicone gel (Experimental): Silicone gel (Kelo-cort™; Advanced Bio-Technologies, Silverdale, WA, USA) From the day of suture removal, the treatment was applied three times daily for 3 months.
  Interventions: Drug: Silicone gel Kelo-cort™;
- Onion extract gel (Active Comparator): Onion extract gel (Contractubex™; Merz Pharma, Frankfurt, Germany) From the day of suture removal, the treatment was applied three times daily for 3 months.
  Interventions: Drug: Onion extract gel Contractubex™
- No treatment (No Intervention): Subjects who assigned In the no treatment group did not receive any topical scar emollients.

INTERVENTIONS:
Drug: Silicone gel Kelo-cort™;
  Arms: Silicone gel
Drug: Onion extract gel Contractubex™
  Arms: Onion extract gel

SUMMARY:
Hypertrophic or keloid scars develop for about 39% to 68% of patients after surgery. The subjective opinion of the patient regarding the scar will often constitute the standard for judging the success or failure of the procedure. Surgical scars are not only a cosmetic concern but they can also cause pain, itching, discomfort, contracture, and other functional impairment. Various treatment options exists for treating hypertrophic scars and keloids, including intralesional steroid injection, dermabrasion, pressure therapy, surgical excision, radiotherapy, cryotherapy, pulse dye, and carbon dioxide laser ablation. However, these treatments often require multiple visits and have limited success. Therefore, prevention and early recognition of hypertrophic scars and keloids are very important in their management.

Among preventive treatments available, silicone gel and onion extract gel have been marketed as products to improve the appearance and texture of surgical scars. Despite its popularity, data demonstrating the efficacy of these gels are lacking. Furthermore, there is no comparative study of silicone gel and onion extract gel for preventing postsurgical hypertrophic or keloid scars. The investigators therefore conducted this randomized controlled trial to compare the efficacy of silicone gel and onion extract gel for the prevention of postsurgical hypertrophic scars. The investigators also compared patient compliance and side effect between two topical gels.

ELIGIBILITY:
Inclusion Criteria:

1. over 18 years of age,
2. Asian,
3. at least 3 cm sized surgical wound in total length,
4. nonpregnant at the time of presentation (i.e., negative for urine pregnancy test or last menstrual period within the last 4 weeks),
5. able to read and write informed consent and questionnaire.

Exclusion Criteria:

1. women who received nearly scar-free surgery such as laparoendoscopic single-site (LESS) surgery or natural orifice transluminal surgery (NOTES);
2. women who developed surgical complications such as wound infection
3. women who had a history of hypertrophic or keloid scarring in abdomen
4. women who were taking chemotherapeutic agents or other medications that would affect wound healing, such as steroids
5. women who had comorbidities such as diabetes, contractive skin disorders (e.g., scleroderma), or active dermatologic conditions
6. women who had allergy to silicone or onion.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2014-02-01 (Actual); Study Completion 2014-05-01 (Actual)

PRIMARY OUTCOMES:
Scar scale (VSS and BIQ) | 3 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- CHA Gangnam Medical Center, Seoul, South Korea